CLINICAL TRIAL: NCT07181044
Title: Effects of Regular Exercise on Ischemia-Modified Albumin and Total Sulfhydryl Levels in Young Women
Brief Title: Exercise, IMA and Sulfhydryl Biomarkers in Young Women
Acronym: IMA-SH & Exerc
Status: Completed | Type: Observational
Sponsor: Duvenciler Anadolu Lİsesi (Other)
Responsible Party: Principal Investigator, Omer Faruk Bilici, Principal Investigator, Duvenciler Anadolu Lİsesi
Other Study IDs: 27750; 27750 (Other: Muş Alparslan University Scientific Research Ethics Committee)
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy Young Women; Regular Exercise; Oxidative Stress; Redox Homeostasis; Antioxidant Defense; Biomarkers; Sports Physiology
Keywords: Ischemia-Modified Albumin; Total Sulfhydryl Groups; Oxidative Stress Biomarkers; Redox Remodeling; Antioxidant Capacity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exercising Women: Healthy women aged 18-25 years who performed structured exercise training ≥3 sessions per week for at least 12 months. Training programs included aerobic, resistance, and flexibility exercise, each session lasting 60-90 minutes.
- Sedentary Controls: Healthy women aged 18-25 years without a history of structured exercise. Physical activity limited to daily living and compulsory school-based physical education classes.

SUMMARY:
Background: Regular physical activity exerts systemic health benefits that extend to redox homeostasis and antioxidant defense mechanisms. Ischemia-modified albumin (IMA) and total sulfhydryl groups (-SH) are increasingly recognized as sensitive biomarkers reflecting oxidative protein modification and thiol-dependent antioxidant capacity, respectively. However, data on their interplay in young women engaged in structured exercise remain scarce.

Objective: This study aimed to investigate the effects of regular exercise on serum IMA and -SH concentrations in healthy young women, thereby providing insights into exercise-induced redox remodeling and sex-specific physiological adaptations.

Methods: A cross-sectional design was employed involving 30 healthy women aged 18-25 years. Participants were divided into an exercise group (n = 15), who had performed structured training ≥3 sessions per week for at least one year, and a control group (n = 15) with no structured exercise history. Venous blood samples were collected after overnight fasting. Serum IMA was quantified using the albumin-cobalt binding assay, and -SH concentrations were determined via the Ellman method. All analyses were performed in duplicate under standardized laboratory conditions. Independent samples t-tests were applied, and effect sizes (Cohen's d) were calculated with 95% confidence intervals.

DETAILED DESCRIPTION:
Regular physical activity is widely recognized as a key determinant of human health, conferring benefits across cardiovascular, metabolic, endocrine, and immune systems. Beyond traditional outcomes, habitual exercise plays a pivotal role in regulating oxidative stress and maintaining redox homeostasis. However, few studies have concurrently investigated ischemia-modified albumin (IMA), a marker of oxidative protein modification, and total sulfhydryl groups (-SH), a marker of thiol-dependent antioxidant defense, particularly in young women. The present study was therefore designed to provide novel insights into exercise-induced redox adaptations in this underrepresented population.

This investigation employed an observational, cross-sectional design conducted in accordance with the STROBE guidelines for reporting observational research. Ethical approval was granted by the Muş Alparslan University Scientific Research Ethics Committee (Approval No: 27750; 01 November 2021), and all procedures complied with the Declaration of Helsinki. Written informed consent was obtained from all participants prior to data collection.

A total of 30 healthy women aged 18-25 years were recruited. Participants were categorized into two groups:

Exercise group (n = 15): Women who had been consistently engaged in structured training for at least 12 months, with a minimum frequency of three sessions per week. Training programs were multimodal and typically included aerobic exercise (e.g., running, cycling, swimming at 60-75% HRmax for 20-30 minutes), resistance training (3 sets of 8-12 repetitions at moderate-to-high intensity, targeting major muscle groups), and flexibility exercises incorporated during warm-up and cool-down phases. Training sessions were supervised by qualified instructors in university or private facilities to ensure adherence to safety standards.

Control group (n = 15): Women without a history of structured exercise, whose activity levels were limited to daily living tasks and compulsory school-based physical education.

Exclusion criteria included chronic cardiovascular, metabolic, or endocrine disorders; smoking or alcohol use; recent use of medications or supplements known to influence oxidative stress; and irregular or intermittent exercise participation. Baseline health screening confirmed all participants were free from chronic illness and suitable for inclusion.

Venous blood samples were collected from the antecubital vein between 07:00 and 09:00 a.m. following an overnight fast of at least 10 hours. Participants refrained from strenuous physical activity, alcohol, and caffeine for 24 hours prior to sampling. Serum was separated by centrifugation and stored at -80 °C until analysis.

Ischemia-modified albumin (IMA): Determined using the albumin-cobalt binding assay (Bar-Or method). Absorbance was measured at 470 nm, expressed in absorbance units (ABSU).

Total sulfhydryl groups (-SH): Measured using the Ellman method, based on the reduction of DTNB and expressed as μmol/L.

All analyses were conducted in duplicate, with strict internal quality control procedures, including calibration curves and reagent blanks. A single trained biochemist blinded to group allocation performed all assays to minimize analytical bias.

Statistical analyses were performed using IBM SPSS Statistics 22.0. Normality was assessed using the Shapiro-Wilk test, and group comparisons were made using independent samples t-tests. Effect sizes (Cohen's d) with 95% confidence intervals were calculated to assess the magnitude of differences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18-25 years
* For exercise group: Regular structured training ≥3 sessions per week for at least 12 months
* For control group: No structured exercise background, only daily living activity

Exclusion Criteria:

* History of chronic cardiovascular, metabolic, or endocrine disorders
* Smoking or alcohol abuse
* Current or recent use (past 6 months) of medications or supplements influencing oxidative stress or hormonal regulation
* Irregular or intermittent exercise participation not meeting the defined threshold

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty healthy women aged 18-25 years were recruited. Fifteen had a history of regular structured exercise training, while fifteen had sedentary lifestyles without structured exercise.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Serum Ischemia-Modified Albumin (IMA) | Baseline (single fasting blood draw)
  Change in serum ischemia-modified albumin (IMA) concentration, measured in absorbance units (ABSU) using the albumin-cobalt binding assay.

SECONDARY OUTCOMES:
Serum Total Sulfhydryl Groups (-SH) | Baseline (single fasting blood draw)
  Change in serum total sulfhydryl (-SH) concentration, measured in μmol/L using the Ellman method.

CONTACTS AND LOCATIONS:
Locations (1):
- Yüzüncü Yıl University, Central Research Laboratory, Van, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involved a small sample of healthy young women and includes sensitive biomarker information. Data sharing is restricted by the ethics committee approval and participant consent, which did not authorize public distribution of individual-level data.

REFERENCES:
- [Derived] Bilici OF, Kahraman MZ, Turker A, Seyhan S, Sahin MF, Demir H, Acar G, Bilici MF, Soylu C, Sogut T, Bakum A. Effects of regular exercise on ischemia-modified albumin and total sulfhydryl levels in young women: a cross-sectional study. Front Physiol. 2025 Nov 20;16:1719454. doi: 10.3389/fphys.2025.1719454. eCollection 2025. PMID 41357165